CLINICAL TRIAL: NCT04534946
Title: A Pilot Study Evaluating the Usability of the Oabi Mobile Application
Acronym: OAB
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Other Study IDs: 2016P002386
Record Dates: First submitted 2018-03-26; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is not an intervention study — This is not an intervention study

SUMMARY:
Our primary purpose is to assess the use feasibility and acceptability of the study phone app called, "Oabi" app with patients diagnosed with overactive bladder disorder (OAB).

DETAILED DESCRIPTION:
Tracking overactive bladder disorder can be an important part of managing the disease. It can help the patient and the health care providers keep a tab on what is working to help manage OAB symptoms. Tracking urination patterns can actually help patients normalize their bladder problems. By focusing on certain behaviors and habits that contribute to their OAB and changing those behaviors, patients can effectively control OAB symptoms. The Oabi mobile application has been created with the goal of helping patients learn more about their day-to-day symptoms as well as track and self-manage their symptoms. Additionally, the Oabi app connects patients with their HCP via a clinician portal to boost communication, and encourage patient-provider interaction. The goal of this pilot study is to evaluate the usability and acceptability of the Oabi mobile app.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of OAB (with active OAB symptoms) with or without urge incontinence who are:

  * Treatment-naive patients who started a new treatment within two weeks prior to the study enrollment
  * Transitioning to another treatment (pharmacotherapy)
  * Transitioning from behavioral therapy to pharmacotherapy
* Adults aged 18 yrs and above.
* Own a Smartphone with Android Operating System with an OS of 5.0 or higher or willing to use a study phone as their primary for the duration of the study (Samsung Galaxy S6).
* Sufficient understanding of the English language to be able to read and understand study procedures.
* Willing to participate in the research study and sign informed consent.
* Has adequate access to the internet to use the app.

Exclusion Criteria:

* Subjects unable or unwilling to participate for at least three months.
* Subjects with vision, hearing, and/or speech problems that may limit their participation in data collection procedures.
* Subjects with physical limitations that limit may their ability to use a Smartphone, effectively navigate a Smartphone app, and type on a Smartphone.
* Participants with the history of urological surgery or those currently using a urinary sling.
* Participants on botox treatment for OAB.
* Participants with OAB symptoms due to coexisting conditions such as urinary tract infection (UTI), and or benign prostatic hypertrophy (BPH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a primary diagnosis of overactive bladder disorder
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Mobile application usability | 12 weeks
  To assess the usability and acceptability of the mobile app via post-pilot survey

SECONDARY OUTCOMES:
User application engagement | 12 weeks
  To assess participant engagement with the Oabi app, to assess provider engagement and satisfaction with the Oabi clinician portal, to assess the perceived value of the app in how it impacts the HCP-patient dialogue and patient care related to the management of OAB (qualitatively), and to gather recommendations for modifications to the Oabi app and clinician portal from users.

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Jethwani, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General/North Shore Center, Salem, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.